CLINICAL TRIAL: NCT04367298
Title: Chronoprevention in Hospital Falls of Older People: A Nursing Intervention CHRONOFALLS
Brief Title: Chronoprevention in Hospital Falls of Older People
Acronym: CHRONOFALLS
Status: Completed | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Andalusian Regional Ministry of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: PI-0360-2017
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Accidental Fall
Keywords: accidental falls; older people; nursing care; nursing; temporal patterns; prevention; circadian rhythms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 34 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronoprevention in hospital falls: Implementation of a hospital preventive measures program: adjusted to the identification of temporal patterns of falls and relative risk factors of falls.
  Interventions: Behavioral: Chronoprevention

INTERVENTIONS:
Behavioral: Chronoprevention — Preventive measures will be focused on organizational, educational and behavioural elements related to older people and healthcare professionals

SUMMARY:
Accidental falls in hospitals are serious events concerning the safety of the patients. Recent studies demonstrated that the time of falls is a key factor to be considered in prevention. It has been shown that the time of day, the day of the week and the month of the year impact on the occurrence of falls.

The aim of this project is to know the effect of the application of a program of preventive measures based on the temporal patterns of the risk factors on the hospital fall occurrence. A mixed method research design will be conducted. Three phases will be carry out: 1) Longitudinal prospective study in two parts: a) audits and seminars of health professionals focused on an effective and efficient hospital falls register. Cosinor and Multi-Component analyses will be performed to obtain temporal patterns of the hospital falls and their related variables. b) Implementation of a based-temporal patterns, multidimensional prevention program. 2) Retrospective study of falls registered in institutional databases. 3) Qualitative study based on focus groups (physicians, nurses and nursing assistants).

It is imperative to study temporal patterns of hospital falls to effectively and comprehensively define the etiology of falls, and therefore, design preventive strategies. A reduction of the number of in-hospital falls and related injuries is expected, as well as, an improvement of the quality of life of patients. Considering temporal patterns, and levels of mood and sleep of healthcare professionals will achieve an improvement of patient safety.

DETAILED DESCRIPTION:
-Design

A mixed-method research will be carried out. Three different study design will be used:

Phase 1. Prospective longitudinal study in 2 steps:

* A first step, of 18 months, in which a first intervention of audits and seminars in health professionals will be carried out, focused on an effective and efficient registry of hospital falls in older people. This first phase is crucial to identify temporal patterns of falls in relation to specific intrinsic and extrinsic risk factors among hospitalized older people; as well as the levels of fatigue/sleepiness, attention and cognitive functionality of the health professionals who attend to an in-hospital fall.
* A second step, of application of a multidimensional prevention program for 15 months focused on organizational, educational and behavioral elements; applied to admitted older people and health professionals.

Phase 2. Retrospective study of the fall records found in the institutional databases of the study centers, in the period between January 2018 - September 2020. This period covers the first (January 2018 - May 2019) and the second phase (June 2019 - September 2020) of the project, previously indicated.

Phase 3. Descriptive exploratory study with a qualitative approach, focus groups made up of health professionals: doctors, nurses and nursing assistants who provide and have provided their professional services in the field of study, in the periods in which the studies have been carried out. longitudinal and retrospective previously mentioned.

ELIGIBILITY:
Inclusion Criteria in patients:

* Patients who suffer a hospital fall
* Accept and sing the informed consent

Exclusion Criteria in patients:

* Do not accept and sign the informed consent

Inclusion Criteria in healthcare professionals:

* Nurses in charge of the care of patients who suffer a fall
* Accept and sing the informed consent

Exclusion Criteria in patients:

* Nurses who do not care for a patient suffering a fall
* Do no accept and sign the informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years who suffer one/several fall/s during their hospital admission to four hospital (one teaching and three non-teaching hospitals)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Participant with Hospital falls | Through study completion, an average of 1 month
  Records of falls coded in the International Classification of Diseases (ICD-10) between codes W00-W19.9

SECONDARY OUTCOMES:
Chronotype of patient | Through study completion, an average of 1 month
  Morningness-Eveningness according to Horne-Östberg Questionnaire (1976). Scores can range from 18-86. Scores of 41 and below indicate "evening types". Scores of 59 and above indicate "morning types". Scores between 42 and 58 indicate "intermediate types".
Quality of life of patient | Through study completion, an average of 1 month
  Short Form 36 Health Survey (SF-36) (Spanish version 2) (Alonso et al. 1996). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
General health status of patient | Through study completion, an average of 1 month
  28-Item General Health Questionnaire (GHQ28) (Spanish version) (Lobo et al. 1985). Scores can range from 0-84. Higher GHQ-28 scores indicate higher levels of distress
Sleep pattern of the healthcare professionals | Through study completion, an average of 1 month
  Pittsburgh Sleep Quality Index (Spanish version) (Macías & Royuela, 1996). Score can range from 0-21 with the higher total score indicating worse sleep quality.
Chronotype of the healthcare professionals | Through study completion, an average of 1 month
  Chronotype according to Horne-Östberg Questionnaire (1976). Scores can range from 18-86. Scores of 41 and below indicate "evening types". Scores of 59 and above indicate "morning types". Scores between 42 and 58 indicate "intermediate types".
Quality of life of the healthcare professionals | Through study completion, an average of 1 month
  Short Form 36 Health Survey (SF-36) (Spanish version 2) (Alonso et al. 1996). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
General health status of the healthcare professional | Through study completion, an average of 1 month
  28-Item General Health Questionnaire (GHQ28) (Spanish version) (Lobo et al. 1985). Scores can range from 0-84. Higher GHQ-28 scores indicate higher levels of distress

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Jesús López Soto, PhD, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba
Locations (1):
- Maimónides Biomedical Research Institute of Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Lopez-Soto PJ, Lopez-Carrasco JC, Fabbian F, Minarro-Del Moral RM, Segura-Ruiz R, Hidalgo-Lopezosa P, Manfredini R, Rodriguez-Borrego MA. Chronoprevention in hospital falls of older people: protocol for a mixed-method study. BMC Nurs. 2021 Jun 6;20(1):88. doi: 10.1186/s12912-021-00618-y. PMID 34092223
- [Derived] Lopez-Soto PJ, Rodriguez-Cortes FJ, Minarro-Del Moral RM, Medina-Valverde MJ, Segura-Ruiz R, Hidalgo-Lopezosa P, Manfredini R, Rodriguez-Borrego MA; CHRONOFALLS project collaborators. CHRONOFALLS: A multicentre nurse-led intervention in the chronoprevention of in-hospital falls in adults. BMC Nurs. 2023 May 5;22(1):149. doi: 10.1186/s12912-023-01322-9. PMID 37143072